CLINICAL TRIAL: NCT05678530
Title: Observational, Non-Interventional Study Supporting Validation of VO2Max Estimation Methods Using Results in Patients Receiving Standard of Care Cardiopulmonary Exercise Tests (CPET)
Status: Recruiting | Type: Observational
Sponsor: Prolaio (Industry)
Responsible Party: Sponsor
Other Study IDs: CTP-020
Record Dates: First submitted 2022-12-05; First posted 2023-01-10 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Cardiopulmonary

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy: Healthy Subjects who undergo the CPET
- Standard of Care: Standard of Care subjects who undergo the CPET as part of routine Standard of Care

SUMMARY:
In this study, the hypothesis being explored is that VO2Max and other CPET parameters can be accurately estimated from biosignals (namely, motion from accelerometers and cardiopulmonary variables from EKG) collected during activities of daily living using wearable biosensors worn by study participants. This study will aim to collect development and validation data for a machine learning algorithm and to evaluate the performance of the algorithm. A total of 1000 participants will be enrolled including: (Normal) 100 participants, self-reported healthy male and female participants aged 18 to 80 and (Standard of Care) 900 participants.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to comply with protocol procedures and available for the duration of the study.
2. Willing to sign and date informed consent document for study participation.
3. Participant is undergoing the Cardiopulmonary Exercise Test (CPET) as Standard of Care

Exclusion Criteria:

1. Participant is pregnant, lactating or ≤30 days post-partum.
2. Participant has limited or no intrinsic sinus node function (i.e. chronic atrial pacing).

   • If participant has an indwelling cardiac device and programming cannot be sufficiently ascertained to assure sinus node competence and lack of atrial pacing, the patient should be excluded.
3. Barostim (™) or similar noncardiac electrical pulse generating device in situ.
4. Complex congenital heart disease (even repaired or palliated) with the following exception:

   • Biventricular physiology without severe valvar dysfunction (e.g. free pulmonary insufficiency) at the discretion of the investigator.
5. Any history of allergy to adhesive
6. Any cognitive or physical limitations that, in the opinion of the investigator, limits the participant's ability to fully follow study procedures and/or reach a respiratory exchange ratio of 1.0.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participant is undergoing the Cardiopulmonary Exercise Test (CPET) as Standard of Care
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-06-06 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Collect development and validation data for a VO2Max (eVO2Max) machine learning algorithm and to evaluate the performance of the algorithm. | March 2025
  Develop an Estimated VO2Max (eVO2Max) algorithm which will estimate a participant's VO2Max value using data collected from physiological wearable biosensors (ECG & Activity).

CONTACTS AND LOCATIONS:
Overall Officials: Greg Kurio, MD, Study Director — Prolaio, Inc
Locations (16):
- United States (15):
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - VA Palo Alto Healthcare System, Palo Alto, California
  - University of California San Francisco, San Francisco, California
  - The Lundquist Institute, Torrance, California
  - Nemours Cardiac Center, Wilmington, Delaware
  - Memorial Healthcare System, Office of Human Research, Hollywood, Florida
  - Mayo Clinic Florida, Jacksonville, Florida
  - New Generation of Medical Research, Naples, Florida
  - physIQ, Chicago, Illinois
  - University of Illinois Hospital & Health Sciences System, Chicago, Illinois
  - Advocate Aurora Health Institute, Oakbrook Terrace, Illinois
  - Mayo Clinic, Rochester, Minnesota
  - Baylor Scott & White Research Institute, Dallas, Texas
  - Baylor Scott & White The Heart Hospital - Plano, Plano, Texas
  - Intermountain Medical Center, Murray, Utah
- Eastern Health Cardiac Rehabilitation, St. John's, Newfoundland and Labrador, Canada

IPD SHARING:
Plan to Share IPD: No